CLINICAL TRIAL: NCT04751435
Title: IMAGINE: IMproving Access to Genetic INformation for Everyone - A Prospective Trial of a Linguistically and Culturally Appropriate Mainstreaming Model for Hereditary Cancer Multigene Panel Testing Among Diverse Cancer Patients
Brief Title: Developing New Educational Materials About Genetic Testing for a Diverse Group of Cancer Patients
Acronym: IMAGINE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-458
Record Dates: First submitted 2021-02-08; First posted 2021-02-12 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Educational Materials for Genetic Testing; Breast Cancer; Ovarian Cancer; Prostate Cancer; Pancreatic Cancer; Colorectal Cancer
Keywords: Educational Materials; Genetic Testing; Hereditary Cancer; Diverse Cancer Patients; Colorectal Cancer; 20-458
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Prostatic Neoplasms; Pancreatic Neoplasms; Colorectal Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cognitive interview intervention for Phase 1 (Experimental): There is no treatment or intervention for Phase 1 of this study. Participants will be asked to participate in a cognitive interview.
  This section will be amended to include the Phase 2 intervention information once the Phase 1 portion of the study is complete. The Phase 1 materials developed, and results obtained, will directly be part of and inform the intervention for Phase 2.Phase 2: participants will be randomized to the standard-of-care arm or the LCAM intervention arm.
  Interventions: Other: Cognitive interview
- Standard of care (Phase II only randomization) (Active Comparator): Participants will receive in-depth pre-test and post-test genetic counseling provided via telegenetics
  Interventions: Behavioral: Standard of care
- LCAM Intervention (Phase II only randomization) (Active Comparator): Participants will receive adapted pretest educational materials from study staff and/or clinical staff and have testing ordered by their oncologist, followed by post-test genetic counseling via telegenetics with a health and genetic "literacy screener" and adapted clinical communication materials.
  Interventions: Behavioral: LCAM intervention

INTERVENTIONS:
Other: Cognitive interview — Researchers will use formative methods to adapt our previously-developed mainstreaming pre-genetic test educational materials plus standard post-test clinical communication materials used by the MSK CGS for use with the diverse patients. Specifically, it will adapt these materials to be responsive to patients' linguistic and literacy needs, and sensitive to their cultural diversity.
  Arms: Cognitive interview intervention for Phase 1
Behavioral: LCAM intervention — Participants will receive adapted pretest educational materials from study staff and/or clinical staff and have testing ordered by their oncologist, followed by post-test genetic counseling via telegenetics with a health and genetic "literacy screener" and adapted clinical communication materials.
  Arms: LCAM Intervention (Phase II only randomization)
Behavioral: Standard of care — Participants will receive in-depth pre-test and post-test genetic counseling provided via telegenetics
  Arms: Standard of care (Phase II only randomization)

SUMMARY:
Genetic testing is a type of test that detects changes to the genes-the DNA instructions that are passed on from the mother and father. The results of a genetic test can confirm whether the participant has a genetic disorder, which is a disease caused in whole or in part by changes to the genes. Genetic testing can also help determine a person's chance of getting or passing on a genetic disorder. Genetic tests use a sample of blood, hair, skin, or other tissue, and they can look at one gene or multiple genes at the same time. Genetic testing may change the options for treating people with certain types of cancer. For example, some medications are more helpful for the treatment of cancer in people with certain gene changes (mutations).

The researchers are doing this study to develop new educational materials about genetic testing for people who speak different languages and have diverse cultural and educational backgrounds. During the study, the staff will interview participants with diverse cultural and educational backgrounds and ask them to review a sample of the educational materials that have been developed so far. Participants will give their opinions on these materials, and the researchers will use participants' feedback to improve the materials.

DETAILED DESCRIPTION:
The objective of this proposal is to develop, test and evaluate a mainstreaming (LCAM) model for hereditary cancer multigene panel testing (MGPT) among many different types of cancer patients. The central hypothesis is that this LCAM genetic testing model will lead to better patient decision-making, psychosocial, and behavioral outcomes than a traditional model of genetic services represented by our standard-of-care arm. In Phase 1, the researchers will first conduct formative research including transcreation and cognitive interviewing to adapt our existing educational materials (brochure and video) and clinical communication materials (clinic visit summary and family dissemination messaging) for the LCAM model to be useful for patients of many different backgrounds. In Phase 2, the researchers will conduct a randomized clinical trial (RCT) to test and evaluate effects of the LCAM model for hereditary cancer MGPT as compared to standard-of-care among the patients treated at local community hospitals. Patients diagnosed with breast, colorectal, ovarian, pancreatic, or prostate cancer will be offered hereditary cancer MGPT through either: i) standard-of-care wherein in-depth pre-test and post-test genetic counseling are provided via telegenetics (videoconferencing), or ii) LCAM intervention wherein patients receive adapted pretest educational materials from study staff and/or clinical staff and have testing ordered by their oncologist, followed by post-test genetic counseling via telegenetics with a health and genetic "literacy screener" and adapted clinical communication materials. Participants will be followed prospectively and will complete assessments consisting of validated and investigator-designed measures. Phase 2 primary outcomes include genetic test decision satisfaction and genetic counseling satisfaction. Secondary outcomes include additional decision-making, psychosocial, and behavioral outcomes.

For Phase 2, participants will be recruited from our partnering sites, which include Kings County Hospital Center, Queens Cancer Center, Jamaica Hospital Medical Center, and the MSK Ralph Lauren Center for Cancer Care. Study staff will identify eligible patients from review of clinic lists and patient medical records, and will also receive direct study referrals from clinicians located at the partnering sites. Study staff will approach eligible patients in order to describe the study, screen them for eligibility (including assessing language proficiency via self-report and prior experience with cancer genetic counseling/testing), and obtain informed consent and collect their contact information.

ELIGIBILITY:
Inclusion Criteria:

Phase 1

* Age ≥ 18 years as per self-report
* Current or previous diagnosis of breast, ovarian, pancreatic, or prostate cancer as per self-report
* Self-identification as Black, Latino, and/or neither Black nor Latino (i.e.,non-Latino, Non black)
* Fluency in English, Haitian Creole, or Spanish as per self-report (for Spanish, we will attempt to recruit a cohort representing a variety of regions where Spanish is spoken, as informed by current data from participating sites, to achieve neutrality in the language) Fluency is defined as an answer of "well" or "very well" on the screening questions for spoken and reading ability.

Phase 2:

* Age ≥ 18 years as per the medical record
* Current or previous diagnosis of breast, colorectal, ovarian, pancreatic, or prostate cancer meeting at least one of the applicable criteria for the cancer type as per the medical record and/or clinician referral:
* Breast cancer criteria:

  * any diagnosis age 65 or younger;
  * diagnosis of triple negative breast cancer at any age;
  * multiple primary breast cancers at any age;
  * under consideration for PARP therapy;
  * any family history (1st, 2nd, or 3rd degree relatives) of ovarian or pancreas cancer, or 1 relative with breast cancer who meets the above criteria, or 2 relatives with breast cancer at any age; or clinician discretion)
* Colorectal cancer criteria:

  * any diagnosis age 50 and below;
  * mismatch repair deficient colorectal cancer;
  * colorectal cancer at any age with an additional Lynch syndromerelated primary cancer at any age;
  * colorectal cancer at any age with a 1st or 2nd degree relative with colorectal cancer at/before age 50;
  * colorectal cancer at any age with 2 or more 1st or 2nd degree relatives with a Lynch syndrome-related cancer at any age
* Ovarian cancer criteria:

  ° invasive ovarian cancer
* Pancreatic cancer criteria:

  ° pancreatic adenocarcinoma
* Prostate cancer criteria:

  * castrate-resistant, metastatic prostate cancer;
  * high-risk prostate cancer (pending pathology definition)
* Fluency in English, Haitian Creole, or Spanish as per self-report. Fluency is defined as an answer of "well" or "very well" on the screening questions for spoken ability
* No prior cancer genetic counseling or germline testing for cancer risk as per self-report clinician's note, and/or no clinical documentation

Exclusion Criteria:

Phase 1:

* Individuals of impaired decision-making capacity as per a clinician's or consenting professional's judgment.
* Subjects who indicate level of fluency as "not at all" or "not well".

Phase 2:

* Individuals of impaired decision-making capacity as per a clinician's or consenting professional's judgment.
* Subjects who indicate level of fluency as "not at all" or "not well".

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 445 (Estimated)
Dates: Start 2021-11-16 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients who complete the cognitive interview (Phase I) | 1 year
  the number of patients who complete the cognitive interview
Genetic test decision (Phase II) satisfaction | 6 months
  is measured with the validated Satisfaction with Decisions scale.
Genetic counseling satisfaction (Phase II) | 6 months
  is measured with the validated Genetic Counseling Satisfaction scale

CONTACTS AND LOCATIONS:
Overall Officials: Jada Hamilton, PhD, MPH, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - Kings County Hopsital Center, Brooklyn, New York
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - Memorial Sloan Kettering at Ralph Lauren Center (Limited Protocol Activities), New York, New York
  - Jamaica Hospital Medical Center (Data Collection Only), Richmond Hill, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm